CLINICAL TRIAL: NCT02907086
Title: Protocol to Permit the Acquisition of Circulating Tumor Material in Colorectal Cancer and Melanoma
Brief Title: Circulating Tumor Material in Colorectal Cancer and Melanoma
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 12916
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer and Melanoma
MeSH Terms: conditions — Colorectal Neoplasms; Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- colorectal cancer
  Interventions: Other: blood collection
- melanoma
  Interventions: Other: blood collection

INTERVENTIONS:
Other: blood collection — Patients will receive a research draw for circulating tumor material analysis with standard clinical labs

SUMMARY:
Observational study to allow the collection of blood and medical information to evaluate the role of circulating tumor material in patients with colorectal cancer and melanoma

ELIGIBILITY:
Inclusion Criteria:

* The subject must be a patient at the Hospital of the University of Pennsylvania

  1. Patients with presumed stage II, III, or IV colorectal cancer with planned surgical resection of either the primary tumor or metastatic lesion(s) being evaluated at the Hospital of the University of Pennsylvania
  2. Patients with histologically confirmed melanoma stage IIb, IIc, IIIa, IIIb, or IIIc/IV scheduled for surgical resection being evaluated at the Hospital of the University of Pennsylvania.
* The subject must be able to provide informed consent or have an acceptable surrogate capable of giving consent on the subject's behalf.
* The subject must be 18 years of age or older.

Exclusion Criteria:

* The subject is not able to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colorectal cancer and melanoma patients
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Number of blood samples collected | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark O'Hara, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States